CLINICAL TRIAL: NCT07284368
Title: Advance Choice Document Implementation
Acronym: ACDI
Status: Enrolling by invitation | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: R&D2025/062; 2946 (Other Grant/Funding Number: Maudsley Charity)
Record Dates: First submitted 2025-11-13; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Detention Under the Mental Health Act
Keywords: Advance Statements; Advance Choice Documents; Psychiatric Advance Directives; Mental Health Act; Involuntary hospitalisation; Coercion; Detention rates

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACD holders: service users with a history of detention under the Mental Health Act that create Advance Choice Documents
  Interventions: Other: Advance Choice Document Implementation

INTERVENTIONS:
Other: Advance Choice Document Implementation — Creation and application of Advance Choice Documents

SUMMARY:
Advance Choice Documents (ACDs) are statements of preferences for mental health care and treatment made when service users have capacity to do so. This is done with their care team and others as desired, e.g. carers/supporters or advocates. In addition to improving therapeutic relationships, ACDs have been shown to reduce compulsory psychiatric admissions by 25%.

South London and Maudsley is currently implementing ACDs into routine practice across its services and the Advance Choice Document Implementation (ACDI) project, run by researchers at King's College London, is supporting the development of related resources and the evaluation of the effectiveness of the implementation. Advisory groups will also guide the study approach throughout.

The project comprises four work packages. Work Package 1 involves focus groups with stakeholders (service users, carers, staff) to inform implementation for Older Adults and CAMHS services. This is to understand the barriers and facilitators for ACD implementation in these services; and learn what adaptations are needed to the ACD resources and procedures for use in these services

Work Package 2 is a prospective study of ACD completion and use throughout all directorates. This will comprise interviews with service users after ACD creation and after an event where the ACD is expected to have been used; interviews with their care-team during expected use events; and interviews/focus groups with staff facilitating the creation of ACDs to understand the integration of their role in SLaM.

Work Package 3 is a retrospective study examining the impact of ACD creation on health service use and routinely collected outcomes. Work Package 4 is a prospective study of ACD use and its relationship to ACD content. Work Packages 3 and 4 will use de-identified data collected via South London an Maudsley's Clinical Records Interactive search System (CRIS).

For more information on ACDI, the people involved, and related publications, please visit: https://www.kcl.ac.uk/research/acdi

ELIGIBILITY:
Inclusion Criteria:

WP1: Focus Groups Service users-Young people Aged ≥ 16 Experienced detention under the MHA while in the care of CAMHS Currently under the care of community mental health services (CAMHS / EI / CMHT)

Older adults

1. Experienced detention under the MHA while under services for Older Adults
2. Currently under the care of older adult community mental health services

Carers / Informal supporters Aged ≥ 16 years A relative or friend of a service user who is eligible for the study

Professionals Professional potentially involved in supporting the completion of ACDs (i.e., community mental health team (CMHT) staff, advocates, peer workers) SLaM professionals potentially involved in referring to ACDs (i.e., inpatient and emergency department liaison mental health staff, home treatment, place of safety and street triage staff) Approved mental health professionals (AMHPs) and Section 12 (MHA) approved doctors involved in detention.

Ambulance, prison mental health and Emergency Department staff General Practitioners, including mental health leads, or other primary care professionals who care for people with SMI discharged from secondary services

WP 2: Prospective study of ACD completion and use Service users All service users: accepted referral to an ACD facilitator for ACD creation Young people

1. Aged ≥ 16
2. Experienced detention under the MHA while in the care of CAMHS
3. Currently under the care of community mental health services (CAMHS / EI / CMHT/)
4. Accepted referral to an ACD facilitator for ACD creation; including participants who decline to complete and ACD after referral to an ACD facilitator.

Older adults

1. Experienced detention under the MHA while under services for Older Adults
2. Currently under the care of older adult community mental health services
3. accepted referral to an ACD facilitator for ACD creation

General Adult:

1. Aged ≥ 18 years
2. Previously detained under the MHA
3. Under the care of community mental health services (CMHT or EI)

Forensic

1. Aged ≥ 18 years
2. Experience detention under the MHA into forensic services
3. Currently under the care of forensic mental health services

Carers: relative or friend of someone referred to an ACD facilitator

Professionals: SLaM staff involved in the care of a participant with an ACD whose ACD is expected to have been consulted because they were: involved in a transfer of care, placed in zoning, referred for a MHA assessment or to a home treatment team, attended an Emergency Department or Place of Safety, admitted to a psychiatric inpatient unit or imprisoned.

The interviews conducted with service users and staff after the expected use event will also include questions about satisfaction with and perceived value of the process of completing, distributing, accessing, honouring, and reviewing an ACD.

Exclusion Criteria:

Service users Aged under 16 years Lacking capacity to provide consent and/or is unwilling to do so Currently detained under the MHA in psychiatric hospital Currently under the care of eating disorder services

Carers/informal supporters Aged under 16 years Is not a relative or friend of a service user who is eligible for the study

Professionals Is not a mental health professional or Section 12 (MHA) approved doctor Is not a professional involved in supporting the completion of ACDs Is not a General Practitioner or mental health lead caring for people with SMI discharged from secondary services.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with severe mental Illnesses
Sampling Method: Non-Probability Sample
Enrollment: 374 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of admissions under the Mental Health Act sections 2, 3, 135 and and associated bed days | 18 months
  Mental Health Act sections Section 2, 3, 135 and 136 are a means to detain someone in a psychiatric facility, in England and Wales.
  Evaluation will be done over different follow-up periods and include participants admitted under all Sections of the Mental Health Act and associated bed-days, compared to number of participants admitted voluntarily (non-Mental Health Act) and associated bed-days.

SECONDARY OUTCOMES:
Number of Home Treatment Team events | 18 months
  The number of Home Treatment Team events and days spent under the care of Home Treatment Teams will be assessed for participants with advance choice documents and those without advance choice documents
Number of events of acute mental health and emergency service use | 18
  The number of events use of acute mental health and emergency services will be evaluated for participants with advance choice documents compared to those without advance choice documents
Rates of restraint | 18
  The number of events where restraint is used will be evaluated for participants advance choice documents compared to participants without advance choice documents, across each follow-up period. As these events are not recorded in structured fields, free-text entries will be searched to identify all events containing the words: Restrained' and/or 'restraint'
Number of days spent in seclusion | 18 months
  The number of days spent in seclusion will be evaluated for participants with advance choice documents compared to those without advance choice documents. As these events are not recorded in structured fields, free-text entries will be searched to identify all events containing the words 'Seclusion' and 'supervised confinement'
Number of events of involuntary medication | 18 months
  The number of events where involuntary medication is used will be evaluated for participants advance choice documents compared to those without advance choice documents
Number of safety events recorded (violence, self-harm, consequences of self-neglect and other serious untoward incidents) | 18 months
  The number of safety events recorded will be evaluated for participants with advance choice documents compared to those without advance choice documents
Number of events of contact with police related to use of mental health services | 18 months
  The number of events of contact with police related to use of mental health services will be evaluated for participants with advance choice documents compared to those without advance choice documents
Number of events of General health service use | 18 months
  General health service use will be measured through data linkage with Hospital Episode Statistics (HES). These data will be obtained at a national level for all service users. Physical health service use outcomes will include: inpatient admissions and associated bed days (this will include Healthcare Resource Group codes, associated primary and secondary diagnostic codes, admission category, and treatment specialty code), Emergency Department (ED) attendances (this will include Healthcare Resource Group codes, diagnosis classifications, investigations codes, treatment codes, arrival mode, and attendance disposal codes), and outpatient appointments (this will include appointment information such as first appointment. We will extract routinely collected outcomes such as the Health of the Nations Outcomes Scales (HoNOS)
Number of community mental health team events | 18 months
  Number of community mental health team events will be evaluated for participants with advance choice documents compared to those without advance choice documents.
Number of psychiatric liaison team events (in emergency departments) | 18 months
  The number of psychiatric liaison team events will be evaluated for participants with advance choice documents and those without. The number of events will be requested for all follow-up periods within 18 months. (ie participants will have varying follow-up periods)

CONTACTS AND LOCATIONS:
Locations (1):
- South London and Maudsley/Institute of Psychiatry, Psychology, and Neuroscience-King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be publicly available due to risk of reidentification.

REFERENCES:
- See also: Related Info — https://www.kcl.ac.uk/research/acdi

DOCUMENTS (2):
  • Study Protocol (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT07284368/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT07284368/SAP_001.pdf